CLINICAL TRIAL: NCT01455896
Title: A Randomized, Multi-Center Study to Evaluate Cardiovascular Outcomes With ITCA 650 in Patients Treated With Standard of Care for Type 2 Diabetes
Brief Title: A Study to Evaluate Cardiovascular Outcomes in Patients With Type 2 Diabetes Treated With ITCA 650
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITCA 650-CLP-107
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ITCA 650 60 mcg/day (Experimental): ITCA 650 is exenatide in DUROS
  Interventions: Drug: ITCA 650
- ITCA placebo (Other)
  Interventions: Other: ITCA placebo

INTERVENTIONS:
Drug: ITCA 650 — ITCA 650
  Arms: ITCA 650 60 mcg/day
Other: ITCA placebo — ITCA placebo
  Arms: ITCA placebo

SUMMARY:
Phase 3 study to Evaluate cardiovascular outcomes in patients with type 2 diabetes treated with ITCA 650.

ELIGIBILITY:
Inclusion Criteria:

* HBA1c > 6.5%
* History of coronary, cerebrovascular or peripheral artery disease

Exclusion Criteria:

* history of pancreatitis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4156 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
time to first occurrence of any event included in the MACE cardiovascular composite endpoint (CV death, non fatal MI, non fatal stroke, or hospitalization for unstable angina), | 2 years

CONTACTS AND LOCATIONS:
Locations (41):
- United States (33):
  - Study Site, Chandler, Arizona
  - Intarcia Therapeutics, Inc, Hayward, California
  - Study Site, Long Beach, California
  - Study Site, Port Hueneme, California
  - Study SIte, San Diego, California
  - Study Site, Bradenton, Florida
  - Study Site, New Port Richey, Florida
  - Study Site, Palm Harbor, Florida
  - Study Site, Chicago, Illinois
  - Study Site, Avon, Indiana
  - Study Site, Evansville, Indiana
  - Study Site, Franklin, Indiana
  - Study Site, Greenfield, Indiana
  - Study Site, Muncie, Indiana
  - Study Site, Newton, Kansas
  - Study Site, Wichita, Kansas
  - Study Site, Metaire, Louisiana
  - Study Site, Rochester, Michigan
  - Study Site, St Louis, Missouri
  - Study Site, Billings, Montana
  - Study Site, Las Vegas, Nevada
  - Las Vegas, Nevada
  - Study Site, Winston-Salem, North Carolina
  - Study Site, Cincinnati, Ohio
  - Study Site, Columbus, Ohio
  - Study Site, Franklin, Ohio
  - Study Site, Pittsburgh, Pennsylvania
  - Study Site, Uniontown, Pennsylvania
  - Study Site, Greer, South Carolina
  - Study Site, Austin, Texas
  - Dallas, Texas
  - Study Site, Dallas, Texas
  - Study Site, San Antonio, Texas
- Plovdiv, Bulgaria
- Hvidovre, Denmark
- Oulu, Finland
- Bad Lauterberg im Harz, Lower Saxony, Germany
- Sopot, Poland
- Martin, Slovakia
- Johannesburg, Gauteng, South Africa
- Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Ruff CT, Baron M, Im K, O'Donoghue ML, Fiedorek FT, Sabatine MS. Subcutaneous infusion of exenatide and cardiovascular outcomes in type 2 diabetes: a non-inferiority randomized controlled trial. Nat Med. 2022 Jan;28(1):89-95. doi: 10.1038/s41591-021-01584-3. Epub 2021 Dec 6. PMID 34873344
- [Derived] Wittbrodt ET, Eudicone JM, Bell KF, Enhoffer DM, Latham K, Green JB. Generalizability of glucagon-like peptide-1 receptor agonist cardiovascular outcome trials enrollment criteria to the US type 2 diabetes population. Am J Manag Care. 2018 Apr;24(8 Suppl):S146-S155. PMID 29693361